CLINICAL TRIAL: NCT05384847
Title: Effects of Triiodothyronine (T3) in Ischemic Heart Failure
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Arshed A. Quyyumi, Professor of Medicine, Emory University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003552
Record Dates: First submitted 2022-04-29; First posted 2022-05-20 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Heart Failure
Keywords: Ischemic Heart Failure; NYHA Class II-III; Implantable Cardioverter Defibrillator (ICD)
MeSH Terms: conditions — Heart Failure | interventions — Triiodothyronine; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Experimental Phase IA (Experimental): In Phase IA two participants (1 and 2) will receive ascending dose levels of the study drug (5 µg T3 orally twice daily for the first 2 days and 10 µg T3 orally twice daily for the next 3 days).
  Interventions: Drug: Thyroid hormone T3
- Experimental Phase IB (Experimental): In Phase IB, dose adjustments will be calculated while accounting for laboratory and safety data from the first two participants (Phase IA) for the remaining 3 participants within the treatment arm of Phase I. Participants 3 to 5 will receive 10 µg T3 orally twice daily on day 1 and 20 µg T3 twice daily from day 2 to 5.
  Interventions: Drug: Thyroid hormone T3
- Control Group-Phase IA and IB (Placebo Comparator): The control group will have testing as the experimental group but will not be given any medications.
  Interventions: Other: Control Group
- Experimental Phase II (Experimental): Patients who were enrolled in the open-label control group of Phase I and who have completed the 3-month follow-up will be permitted to enroll in Phase II. This Phase will start treatment after completion of Phase I and approval from the Data and Safety Monitoring Board (DSMB) to proceed with a single cohort that will receive a stable dose of the study drug (20 µg T3 orally twice daily for 5 days).
  Interventions: Drug: Thyroid hormone T3

INTERVENTIONS:
Drug: Thyroid hormone T3 — Participants will be admitted to the General Clinical Research Center (GCRC) for up to 5 days and will receive study medication twice a day. Participants will receive oral T3 under the supervision of the Principal Investigator or qualified co-investigators at the GCRC. The study drug will be given within 30 days after enrollment.
  Other Names: Triiodothyronine; Cytomel
  Arms: Experimental Phase IA; Experimental Phase IB; Experimental Phase II
Other: Control Group — The control group will have testing and study procedures as per protocol but will not be admitted to the General Clinical Research Center (GCRC) and will not receive the study medication. After completion of phase I, participants will be permitted to enroll in Phase II.
  Other Names: No intervention
  Arms: Control Group-Phase IA and IB

SUMMARY:
This study aims to determine whether giving triiodothyronine (T3), a thyroid hormone, is safe and helps improve symptoms and signs of heart failure.

The study is divided into 2 phases. In the first phase, participants have a 50-50 chance of receiving the study drug. Participants who are enrolled to receive the study drug will be admitted to the General Clinical Research Center (GCRC) for 5 days for oral thyroid hormone treatment and monitoring. They will have 4 additional follow-up visits over the next year. Participants who are not enrolled to receive the study drug will not be admitted but will have similar follow-up visits in the outpatient setting. Participants who do not receive the drug in Phase I will have the opportunity to enroll in Phase II of the study where everyone will receive the thyroid hormone treatment.

If this study finds that patients have improved heart function after treatment with thyroid hormone without unacceptable side effects, this could result in a new treatment for patients with heart failure.

DETAILED DESCRIPTION:
About six million adults in the United States have heart failure (HF). Myocardial ischemic injury is the most common trigger of HF and most deaths after a myocardial infarction (MI) are preceded by HF. Treatment for HF with reduced ejection fraction (HFrEF) consists of beta-adrenergic receptor antagonists, antagonists of the renin-angiotensin-aldosterone system (ACEI, ARB, angiotensin receptor neprilysin inhibition), aldosterone antagonists, and Sodium-glucose Cotransporter-2 (SGLT-2) antagonists. Despite these guideline-directed therapies, 1 in 2 HF patients dies within 5 years of diagnosis, a death rate similar to that of some cancers. Thus, the development of next-generation therapies to treat HF represents an important unmet clinical need.

The overarching goal of these preclinical and anticipated clinical studies is to develop translatable strategies, using transient triiodothyronine (thyroid hormone T3) administration in patients with HF receiving beta1-adrenergic receptor (AR) blocker therapy (metoprolol succinate) with other HF medications, to permanently improve left ventricular (LV) contractile function by regenerating cardiac muscle.

The most-cited basis of ineffective cardiac regeneration in mammals is the low proliferative capacity of adult cardiomyocytes. The investigators have sought to understand the most important aspects of these processes to develop therapies that can be used to build or rebuild heart muscle in diseased hearts.

In brief, the investigators' preclinical studies show that T3+metoprolol therapy regenerates heart muscle by increasing cardiomyocytes around the scar and increases the left ventricular ejection fraction (LVEF) thereby restoring LV wall contractility in the scar region. De novo cardiomyogenesis requires neovascularization along with cardiomyocyte proliferation so that the nutrient and oxygen demands of the expanding myocardium are met. Our preliminary studies also show that in chronic post-MI hearts, the mid-apical LV myocardium was repopulated with cardiomyocytes following T3+metoprolol therapy and, in this myocardium, cardiomyocytes were not hypertrophied (data not shown). Importantly, the researchers found no significant differences in mid-apical capillary-to-cardiomyocyte ratios between T3+metoprolol treated post-MI hearts and uninjured age-matched controls.

Together, these findings suggest lasting regenerative repair of hearts with severe preexisting ischemic injury after a brief period of T3+metoprolol combination therapy. Importantly, over the course of this 5-month follow up the research team did not observe any signs of arrhythmias or increase in mortality in mice treated with T3+metoprolol combination therapy. Low free T3 levels (<2.5pg/ml) are found in approximately 10% of patients with early HF and 58% of patients with late HF and are more frequently observed in patients with HF of NYHA class III-IV. This is likely secondary to the upregulation of type 3 iodothyronine deiodinase. Low T3 levels correlate with LVEF and BNP levels in HF. Importantly, a low T3 level in addition to BNP levels is an independent predictor of worse outcomes in patients with HF and after MI. The T3 production rate in normal humans is 16 ± 3 μg/m2 BSA/day. In patients with HF and low T3 levels, 20 μg/m2 BSA/d T3 increased T3 levels significantly to within the normal range. The rate of infusion on days 2 and 3 was then lowered to 13.4 μg/m2 BSA/day on average to maintain this level. There was a concomitant decrease in T4 (10.9 to 9.6 pg/ml) and thyroid-stimulating hormone (TSH) from 2.43 to 0.55 IU but they remained in the normal range.

Based on previous experience in patients with HF, researchers propose to employ a 5-day oral treatment with L-T3 in gradually increasing doses to rapidly establish higher T3 levels in patients with stable ischemic HF with an EF≤40%. The team anticipates that doses of T3 used in the proposed studies will not cause tachycardia or dysrhythmias. Even though the final L-T3 dose proposed here is twice that was previously used, the team believes that the possibility of inducing tachycardia is likely to be low because of the concomitant treatment with metoprolol succinate, a B1-selective (cardioselective) adrenergic receptor blocker therapy. Researchers do not anticipate the development of other hyperthyroid symptoms in these patients as L-T3 administration is only for a brief period of 5 days.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-80 years, male or female;
* Confirmed diagnosis of ischemic HF with left ventricular ejection fraction (LVEF) ≤ 40% (measured by echocardiography within 1 month of Screening);
* Stable symptoms; NYHA class II-III without recent admission (1 month) for acute decompensation;
* Receiving guideline-based standard HF therapies at the maximum tolerated doses for >1 month. Patients on other beta-blockers will be switched to metoprolol succinate at equivalent doses for 3 weeks.
* Presence of ICD for >1 month or implantable cardiac resynchronization therapy defibrillator (CRT-D) for >3 months
* Understand and sign the informed consent form.

Exclusion Criteria:

* LVEF > 40%;
* Unremitting atrial fibrillation during the screening period or clinically significant ventricular tachycardia (on ICD interrogation);
* Non-ischemic HF including hypertrophic cardiomyopathy, peripartum or chemotherapy-induced cardiomyopathy, other non-ischemic cardiomyopathies, constrictive pericarditis, significant and uncorrected valvular heart disease (severe regurgitation or severe stenosis or valvular disease requiring surgery), congenital heart disease, primary pulmonary hypertension or secondary severe pulmonary hypertension (≥ 70 mmHg); large pericardial or pleural effusions; right heart failure due to lung disease;
* Recent admission (1 month) for acute decompensated HF;
* Angina pectoris, cerebrovascular accident, myocardial infarction, revascularization (PCI or other surgery), carotid artery or other large vessel surgery, or cardiac resynchronization therapy (CRT) implant within the past 3 months;
* Planned revascularization within 6 months;
* History of heart transplantation, use of ventricular assist device (VAD) or preparation for heart transplantation, VAD;
* Liver dysfunction (bilirubin or alkaline phosphatase > 2 times the upper limit of normal (ULN), aspartate aminotransferase or alanine aminotransferase > 3 times the upper limit of normal), estimated glomerular filtration rate (eGFR) calculated using the Modification of Diet in Renal Disease Study (MDRD) method < 30 ml/min/1.73 m2;
* Systolic blood pressure < 90 mmHg or > 160 mmHg;
* Blood K+ < 3.2 mmol/L or > 5.5 mmol/L;
* Women of childbearing age who are planning to become pregnant within 2 years, and pregnant or lactating women;
* Patients whose survival time is expected to be less than 6 months as judged by the investigator;
* Those who have participated in any drug clinical trial within the previous 3 months;
* Severe neurological disorders (Alzheimer's disease, progressive parkinsonism);
* The subjects with a history of cancer that limits life expectancy to <1 year;
* Endocrine disorders include thyroid disease, thyroid replacement therapy, pheochromocytoma, thyromegaly, etc.
* The subject, in the judgment of the Investigator, is unable to complete the study or to comply with the requirements of the study (for administrative or other reasons);
* Prisoners;
* Adults unable to consent;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-12-02 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Changes in the presence of clinical arrhythmias | Baseline, Days 1*, 2*, 3*, 4*, 5*, 6 weeks, 3 months, 6 months, 12 months
  An electrocardiogram will be performed during each study visit and the presence of any Clinical arrhythmias such as ectopy, atrial fibrillation, ventricular arrhythmias, ICD firing will be documented. *Days 1 through 5 apply only to those who are admitted to the GCRC unit.
The number of participants with Angina, acute coronary syndrome, death during the first week | During the first week of treatment period
  The total number of subject's events during the first week of the treatment period will be recorded

SECONDARY OUTCOMES:
Change in left ventricular ejection fraction (LVEF) | Baseline, Day 45, Day 90
  An echocardiogram will be performed at specific study visits and LVEF will be measured
Change in 6-minute walk distance (6MWD) | Baseline, Day 45, Day 90
  Two 6-minute walk tests will be completed at least 2 hours apart to establish a baseline. The mean of the 2 distances will be used as the baseline. The six-minute walk test requires a 100-ft hallway. This test measures the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes. The six-minute walk test serves as a standardized test for functional capacity quantification of HF patients and is predictive of adverse cardiovascular outcomes. Most patients do not achieve maximal exercise capacity during the 6-minute walk test; instead, they choose their own intensity of exercise and can stop and rest during the test.
Changes in New York Heart Association (NYHA) classification | Baseline, Day 45, Day 90
  Participants will be asked about exertional symptoms for NYHA functional categorization of HF symptoms at all time points. Symptom-based scores range from I to IV. The NYHA classification system also includes an objective assessment of cardiovascular disease severity, which ranges from A-D. Differences between treatment and control arms over time will be analyzed as well as within arms over time.
Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) | Baseline, Day 45, Day 90
  This is a disease-specific health status instrument composed of 23 items that quantify the domains of physical limitation, symptoms, self-efficacy, social limitation, and quality of life limitation due to HF. Scores range from 0 to 100. For the KCCQ overall summary score, a small but clinically meaningful change is ≥ 5 points.
Changes in Brain natriuretic peptide (BNP) levels | Baseline, Day 45, Day 90
  -B-type natriuretic peptide (BNP) will be measured at specific study visits. Differences between treatment and control arms over time will be analyzed as well as within arms over time.

OTHER OUTCOMES:
Changes in the Left ventricular end-systolic volume (LVESV) and Left ventricular end-diastolic volume (LVEDV) | Baseline, Day 45, Day 90
  An echocardiogram will be performed at specific study visits and LVESV and LVEDV will be measured.
Changes Left ventricular end-systolic volume index (LVESVI) and end-diastolic volume index (LVEDVI) | Baseline, Day 45, Day 90
  An echocardiogram will be performed at specific study visits and LVESVI and LVEDVI will be measured.
Changes in the LV posterior wall (LVPW) thickness by speckle-tracking echocardiography | Baseline, Day 45, Day 90
  An echocardiogram will be performed at specific study visits where the LV posterior wall (LVPW) thickness by 2D echocardiography (longitudinal and circumferential strain and strain rate).
Changes in longitudinal and circumferential strain by speckle-tracking echocardiography | Baseline, Day 45, Day 90
  An echocardiogram will be performed at specific study visits where longitudinal and circumferential strain will be measured by 2D echocardiography (and strain rate).
Changes in the strain rate by speckle-tracking echocardiography | Baseline, Day 45, Day 90
  An echocardiogram will be performed at specific study visits where the strain rate will be measured by 2D echocardiography
Composite of all-cause mortality | After 1 week of study drug administration up to 12 months
  The total number of subject deaths after the first week of treatment up to 12 months will be recorded
Number of participants with hospital admission due to acute coronary syndrome (ACS) and all-cause HF admissions after first week | After 1 week of study drug administration up to 12 months
  Participants will be asked about any ACS and HF hospital admission during each study visit, in addition, electronic medical records (EMR) will be reviewed periodically to document any ACS and HF hospital admission.

CONTACTS AND LOCATIONS:
Overall Officials: Arshed A. Quyyumi, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital (EUH), Atlanta, Georgia
  - Emory University Hospital Clinical Research Network, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No